CLINICAL TRIAL: NCT02953405
Title: Prescription and Persistence of Antithrombotic Agents in Acute Ischemic Stroke or Transient Ischemic Attack Patients With MCA(Middle Cerebral Artery) Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_CLO001
Record Dates: First submitted 2016-10-25; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: MCA - Middle Cerebral Artery Dissection
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Clopidogrel

SUMMARY:
Prescription and Persistence of Antithrombotic agents in Acute Ischemic Stroke or Transient Ischemic Attack Patients with MCA(Middle Cerebral Artery) Disease.

ELIGIBILITY:
Inclusion Criteria:

* 19 years later, men and women

Exclusion Criteria:

* Subject who is judged to be ineligible by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prescription and Persistence of Antithrombotic Agents in Acute Ischemic Stroke or Transient Ischemic Attack Patients With MCA(Middle Cerebral Artery) Disease
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Prescription status of Antithrombotic Agents | at 12 months after baseline(onset)

CONTACTS AND LOCATIONS:
Locations (1):
- SNUBH, Seoul, South Korea